CLINICAL TRIAL: NCT02920957
Title: Performance Comparison Between Comfilcon A and Senofilcon C Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-70
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- comfilcon A (Active Comparator): Participants are randomized to wear the comfilcon A lens for one month during the cross over study.
  Interventions: Device: comfilcon A
- senofilcon C (Active Comparator): Participants are randomized to wear the senofilcon C lens for one month during the cross over study.
  Interventions: Device: senofilcon C

INTERVENTIONS:
Device: comfilcon A — contact lens
  Arms: comfilcon A
Device: senofilcon C — contact lens
  Arms: senofilcon C

SUMMARY:
The aim of this study is to determine the clinical performance of comfilcon A in comparison to senofilcon C.

DETAILED DESCRIPTION:
This is a prospective, multi-center, bilateral, double-masked, randomized, cross-over, daily wear, two month dispensing study comparing the clinical performance of comfilcon A and senofilcon C lenses after one month of wear.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 34 years of age (inclusive)
* Has had a self-reported eye exam in the last two years
* Is a spherical soft contact lens wearer
* Has a contact lens spherical prescription between -1.00 to -6.00 (inclusive)
* Has a spectacle cylinder no greater than 0.75D (Diopters) in each eye.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Has a contact lens prescription that fits within the available parameters of the study lenses.
* Is willing and anticipated to be able to comply with the wear schedule (at least 6 days per week, 12 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has a history of not achieving comfortable CL (contact lens) wear (defined as 6 days per week; > 10 hours/day)
* Presents with clinically significant anterior segment abnormalities
* Presents with ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Presents with slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Significant pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (or history in past year)
  * Seborrheic eczema of eyelid region, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.
* Is habitually using rewetting/ lubricating eye drops more than once per day
* Is currently wearing daily disposable lenses

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11-23 (Actual); Study Completion 2016-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FAAO, FIACLE, FBCLA, Study Director — Centre for Contact Lens Research
Locations (5):
- United States (5):
  - Golden Optometric Group, Whittier, California
  - Coan Eye Care & Optical Boutique, Ocoee, Florida
  - Cornea & Contact Lens Institute of Minnesota, Edina, Minnesota
  - Sacco Eye Group, Vestal, New York
  - Vision Professionals, New Albany, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 88 participants enrolled for this study, with 1 participant failed the screening leading to 87 who were fitted with and dispensed contact lenses.
Groups:
- Comfilcon A First Then Senofilcon C: Participants randomized to wear the comfilcon A lens first then crossover to Senofilcon C
- Senofilcon C First Then Comfilcon A: Participants randomized to wear the senofilcon C lens first then crossover to comfilcon A
Period: First Intervention : 1 Month
Arm/Group | Comfilcon A First Then Senofilcon C | Senofilcon C First Then Comfilcon A
Started | 46 | 41
Completed | 42 | 41
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Second Intervention: 1 Month
Arm/Group | Comfilcon A First Then Senofilcon C | Senofilcon C First Then Comfilcon A
Started | 42 | 41
Completed | 42 | 40
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Entire Study Population
Groups:
- Overall Baseline Characteristics: Includes groups randomized to wear comfilcon A lens first and senofilcon C lens first.
Arm/Group | Overall Baseline Characteristics
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 27.9 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Lens Fit Acceptance
Description: Investigator fit acceptability for comfilcon A and senofilcon C lenses. Scale 0-4, 0=should not be worn, 1=borderline but unacceptable, 2=minimally acceptable, early review, 3=not perfect but OK to dispense, 4=perfect.
Time Frame: Up to 1 month
Population: Analysis numbers differ from baseline due to protocol deviation and exclusion of subjects lost after only 1 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A at Dispense; Comfilcon A After 2 Weeks; Comfilcon A After 1 Month: Participants are randomized to wear the comfilcon A lens for one month either as the first or second intervention.
  comfilcon A: contact lens
- Senofilcon C at Dispense; Senofilcon C After 2 Weeks; Senofilcon C After 1 Month: Participants are randomized to wear the senofilcon C lens for one month either as the first or second intervention.
  senofilcon C: contact lens
Arm/Group | Comfilcon A at Dispense | Comfilcon A After 2 Weeks | Comfilcon A After 1 Month | Senofilcon C at Dispense | Senofilcon C After 2 Weeks | Senofilcon C After 1 Month
Number analyzed (Participants) | 85 | 84 | 82 | 83 | 82 | 83
units on a scale | 3.6 (0.5) | 3.5 (0.6) | 3.5 (0.7) | 3.5 (0.7) | 3.5 (0.6) | 3.3 (0.8)

2. Primary Outcome: Corneal Coverage
Description: Corneal coverage for comfilcon A and senofilcon C lenses. (yes/no)
Time Frame: Up to 1 month
Population: Analysis numbers differ from baseline due to protocol deviation and exclusion of subjects lost after only 1 visit.
Measure: Number; unit: participants
Groups:
- Comfilcon A at Dispense; Comfilcon A After 2 Weeks; Comfilcon A After 1 Month: Participants are randomized to wear the comfilcon A lens for one month either as the first or second intervention.
- Senofilcon C at Dispense; Senofilcon C After 2 Weeks; Senofilcon C After 1 Month: Participants are randomized to wear the senofilcon C lens for one month either as the first or second intervention.
Arm/Group | Comfilcon A at Dispense | Comfilcon A After 2 Weeks | Comfilcon A After 1 Month | Senofilcon C at Dispense | Senofilcon C After 2 Weeks | Senofilcon C After 1 Month
Number analyzed (Participants) | 85 | 84 | 82 | 83 | 82 | 83
participants
  Yes | 85 | 84 | 82 | 83 | 82 | 83
  No | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Lens Centration
Description: Lens centration for comfilcon A and senofilcon C lenses. (optimum/ decentration acceptable/ decentration unacceptable)
Time Frame: Up to 1 month
Population: Analysis numbers differ from baseline due to protocol deviation and exclusion of subjects lost after only 1 visit.
Measure: Number; unit: participants
Arm/Group | Comfilcon A at Dispense | Comfilcon A After 2 Weeks | Comfilcon A After 1 Month | Senofilcon C at Dispense | Senofilcon C After 2 Weeks | Senofilcon C After 1 Month
Number analyzed (Participants) | 85 | 84 | 82 | 83 | 82 | 83
participants
  Optimum | 77 | 78 | 76 | 71 | 71 | 76
  Acceptable | 7 | 6 | 5 | 11 | 10 | 5
  Unacceptable | 1 | 0 | 1 | 1 | 1 | 2

4. Primary Outcome: Post-blink Movement
Description: Post-blink movement for comfilcon A and senofilcon C lenses. Scale 0-4, (1 step size) (0=Insufficient, 4=Excessive, unacceptable movement)
Time Frame: Up to 1 month
Population: Analysis numbers differ from baseline due to protocol deviation and exclusion of subjects lost after only 1 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A at Dispense | Comfilcon A After 2 Weeks | Comfilcon A After 1 Month | Senofilcon C at Dispense | Senofilcon C After 2 Weeks | Senofilcon C After 1 Month
Number analyzed (Participants) | 85 | 84 | 82 | 83 | 82 | 83
units on a scale | 1.8 (0.5) | 1.9 (0.5) | 1.9 (0.5) | 1.9 (0.6) | 1.9 (0.4) | 1.8 (0.6)

5. Primary Outcome: Lens Lag at Primary Gaze
Description: Lens lag at primary gaze for comfilcon A and senofilcon C lenses. (mm, 0.1 step size)
Time Frame: Up to 1 month
Population: Analysis numbers differ from baseline due to protocol deviation and exclusion of subjects lost after only 1 visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Comfilcon A at Dispense | Comfilcon A After 2 Weeks | Comfilcon A After 1 Month | Senofilcon C at Dispense | Senofilcon C After 2 Weeks | Senofilcon C After 1 Month
Number analyzed (Participants) | 85 | 84 | 82 | 83 | 82 | 83
millimeters | 0.2 (0.2) | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1)

6. Primary Outcome: Tightness on Push up
Description: Tightness on push up for comfilcon A and senofilcon C lenses. Scale 0%-100%, 0%=falls from cornea, 50%=optimum, 100%=no movement)
Time Frame: Up to 1 month
Population: Analysis numbers differ from baseline due to protocol deviation and exclusion of subjects lost after only 1 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A at Dispense | Comfilcon A After 2 Weeks | Comfilcon A After 1 Month | Senofilcon C at Dispense | Senofilcon c After 2 Weeks | Senofilcon C After 1 Month
Number analyzed (Participants) | 85 | 84 | 82 | 83 | 82 | 83
units on a scale | 54 (10) | 51 (9) | 51 (8) | 54 (9) | 53 (9) | 53 (9)

7. Primary Outcome: Lens Wettability
Description: Lens wettability for comfilcon A and senofilcon C lenses. Scale 0-4, (0.5 step size) (0=very poor, 4=excellent)
Time Frame: Up to 1 month
Population: Analysis numbers differ from baseline due to protocol deviation and exclusion of subjects lost after only 1 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A at Dispense | Comfilcon A After 2 Weeks | Comfilcon A After 1 Month | Senofilcon C at Dispense | Senofilcon C After 2 Weeks | Senofilcon C After 1 Month
Number analyzed (Participants) | 85 | 84 | 82 | 83 | 82 | 83
units on a scale | 3.8 (0.4) | 3.5 (0.6) | 3.4 (0.8) | 3.7 (0.4) | 3.3 (0.7) | 3.3 (0.6)

8. Primary Outcome: Deposit Grading
Description: Deposit grading for comfilcon A and senofilcon C lenses. Scale 0-4 (0.5 step size) (0=no deposits, 4=severe deposits)
Time Frame: Up to 1 month
Population: Analysis numbers differ from baseline due to protocol deviation and exclusion of subjects lost after only 1 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A at Dispense | Comfilcon A After 2 Weeks | Comfilcon A After 1 Month | Senofilcon C at Dispense | Senofilcon C After 2 Weeks | Senofilcon C After 1 Month
Number analyzed (Participants) | 85 | 84 | 82 | 83 | 82 | 83
units on a scale | 0.0 (0.2) | 0.3 (0.6) | 0.5 (0.7) | 0.1 (0.3) | 0.4 (0.7) | 0.7 (0.8)

ADVERSE EVENTS:
Description: Assessment of adverse events was performed during the study visits. Investigators may be notified of adverse events by the participants outside of the study visits.
Groups:
- Comfilcon A: Participants are randomized to wear the comfilcon A lens for one month during either as the first or second intervention.
- Senofilcon C: Participants are randomized to wear the senofilcon C lens for one month during either as the first or second intervention.
Arm/Group | Comfilcon A | Senofilcon C
Serious Adverse Events (participants affected / at risk) | 1/87 | 0/83
Other Adverse Events (participants affected / at risk) | 0/87 | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comfilcon A (N=87) | Senofilcon C (N=83)
Motocycle Accident (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any results communications and has ability to review.